CLINICAL TRIAL: NCT00204126
Title: Determination of Novel Methods of Exercise Testing During Treadmill Gait in Incomplete Spinal Cord Injury
Brief Title: Exercise Testing During Treadmill Gait in Incomplete Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: GUTreadmillSCI
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Spinal Cord Injury
Keywords: exercise testing; treadmill; incomplete spinal cord injury; novel methods
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Device: Treadmill with partial body weight support
Device: Surface Functional Electrical Stimulation

SUMMARY:
Treadmill therapy has the potential to improve the physical fitness and voluntary function of incomplete-lesion spinal cord injured (SCI) patients. However, if it is to be offered as a rehabilitation strategy, evidence must be gathered to support its effectiveness. Present methods used to determine the efficacy of treadmill training do not provide accurate means of monitoring changes in physical fitness during the exercise, or to accurately measure the changes in voluntary muscle function which may occur during a training intervention.

We are therefore currently recruiting subjects for a study investigating the feasibility of new methods for monitoring improvements in physical fitness during walking on a treadmill. We also aim to develop methods for monitoring changes in voluntary muscle strength. The bone density of both legs will also be measured to determine if any improvement has occurred following training.

DETAILED DESCRIPTION:
Treadmill therapy has the potential to improve the cardiopulmonary fitness, voluntary function, and lower limb bone density of incomplete spinal cord injury (SCI) patients. However, if it is to be offered clinically as a rehabilitation strategy then evidence must be gathered to support its effectiveness.

The efficacy of FES-assisted walking with incomplete SCI individuals, both overground and on a treadmill, has previously been assessed by monitoring walking speed, stride length, endurance, cadence, the physiological and oxygen cost, % body weight support (treadmill), and by performing observational gait analysis and manual muscle testing (1,2,3,4,5,6). However, these methods do not provide a means of measuring changes in fitness or for accurately monitoring improvements in voluntary muscle function.

At present appropriate methods for testing a person's cardiopulmonary fitness on a treadmill are lacking. Previously, incremental exercise tests have been carried out by maintaining a constant inclination and increasing the speed linearly.

However, if the speed is increased linearly it is likely that it will increase at too fast a pace. Therefore the test will become a measure of the subject's ability to move their legs quickly and/or efficiently enough, rather than metabolic factors. If a steep gradient is chosen as the constant inclination then a high initial metabolic cost will result, which will limit the test time. Another common method used is to maintain a constant speed while increasing the sine of the angle of inclination. The problem with this method of testing is that if too low a speed is selected then a very steep gradient results before the level of tolerance is reached, and if too high a speed is selected there is a high initial metabolic cost. These problems were addressed in a recent paper by Porszasz et al., 2003 (7). They demonstrated that by increasing walking speed linearly and treadmill gradient curvilinearly, a linear increase in work rate occurs with the subjects fatiguing at a moderate speed. If this protocol could be adapted for use with incomplete SCI patients it would provide an accurate means of testing changes in cardiopulmonary function which may result after treadmill training.

It has recently been recorded that dynamometry (rather than manual muscle scores) should be used to assess changes in voluntary function in incomplete SCI patients (8). Therefore we will employ this approach in this study. Following a spinal injury there is a rapid decline in bone mineral density which increases the risk of fracture following minor trauma. Therefore we will also measure the bone density at the epiphyses and shaft of the tibia and femur to determine if this form of training leads to changes in bone mineral density in this patient population.

By demonstrating that treadmill training can improve the cardiopulmonary fitness of individuals with incomplete SCI, their voluntary strength, and bone mineral density, it will help to provide the evidence that this form of rehabilitation is worthwhile.

By increasing cardiopulmonary fitness it will reduce their risk of developing cardiovascular disease, a major problem in this population due to their sedentary lifestyle. If it can be demonstrated to improve their voluntary function it would suggest that their quality of life and ability to carry out activities of daily living may also improve. Improving their bone density would consequently reduce their risk of fracture. Therefore the results of this study will contribute to the quest of trying to improve the overall health and functional ability of this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory general medical examination
* Incomplete paraplegia or tetraplegia secondary to spinal cord lesion
* Previously discharged from hospital, following primary rehabilitation
* Capable of independent ambulation, with or without orthotic support

Exclusion Criteria:

* Female subjects should not be pregnant.
* No significant history of autonomic dysreflexia.
* No history of significant osteoporosis, or associated previous history of spontaneous lower-limb fracture. Bone density will be measured in the epiphyses of the tibia and femur of both legs using peripheral Quantitative Computed Tomography (pQCT).
* No history of coronary heart disease.
* No clinical features of significant cardio-respiratory impairment.
* Absence of hypertension.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 4
Dates: Start 2005-02; Study Completion 2005-02

PRIMARY OUTCOMES:
peak oxygen uptake
lactate threshold
oxygen uptake kinetics

SECONDARY OUTCOMES:
torque during maximum voluntary contractions in leg muscles
central activation ratio of leg muscles
bone mineral density in tibia and femur

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Hunt, BSc, PhD, DSc, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - University of Glasgow, Glasgow, Lanarkshire
  - Queen Elizabeth National Spinal Injuries Unit, Glasgow, Lanarkshire

REFERENCES:
- [Background] Granat M, Keating JF, Smith AC, Delargy M, Andrews BJ. The use of functional electrical stimulation to assist gait in patients with incomplete spinal cord injury. Disabil Rehabil. 1992 Apr-Jun;14(2):93-7. doi: 10.3109/09638289209167078. PMID 1600188
- [Background] Porszasz J, Casaburi R, Somfay A, Woodhouse LJ, Whipp BJ. A treadmill ramp protocol using simultaneous changes in speed and grade. Med Sci Sports Exerc. 2003 Sep;35(9):1596-603. doi: 10.1249/01.MSS.0000084593.56786.DA. PMID 12972882